CLINICAL TRIAL: NCT03115164
Title: Astrocytoma / Desmoplastic Gamliogliomes (DIA / DIG) - Study of the French Cohort of the Last 20 Years : Clinical, Anatomopathological, Molecular and Radiological Charactersics
Acronym: DIA/DIG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0030
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Astrocytoma; Ganglioglioma Desmoplastics and Infantile
MeSH Terms: conditions — Astrocytoma | interventions — 4-(4-dihexadecylaminostyryl)-N-methylpyridium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with DIA / DIG treated at the French SFCE pediatric
  Interventions: Other: To study the characteristics of patients with DIA / DIG

INTERVENTIONS:
Other: To study the characteristics of patients with DIA / DIG — Describe the characteristics of patients with DIA / DIG treated in French SFCE pediatric oncology centers according to whether these tumors behave in a benign or malignant manner.

SUMMARY:
Astrocytomas / infantile desmoplastic gangliogliomas (DIA / DIG) are rare brain tumors usually affecting infants. They represent about 0.5% of all pediatric brain tumors. DIA / DIG occurs mainly in the first 2 years of life, with a sex ratio M / F of 1.7 to 1. From a histological point of view, DIA / DIG are neuroepithelial tumors. These tumors may have a purely astrocytic differentiation (DIA) or be composed of tumor cells with astrocytic and neuronal differentiation (DIG). The desmoplastic component is usually adjacent to the meninges and is defined by the increase or modification of connective tissues related to the presence of neoplastic cells with the formation of a collagen-rich extracellular matrix.

Due to their benign biological behavior and favorable clinical course, they are classified in benign tumors, ie grade I according to the WHO classification. However, all tumors called DIA / DIG do not behave in a benign manner. Cases of metastatic cerebrospinal and malignant disorders have been described. It appears that about 40% of DIG cases require additional medical treatment such as chemotherapy, radiotherapy and / or new surgery, and 15% of infants and children with GIDD die from the disease. It is possible that what is grouped within the DIA / DIG is a heterogeneous group of tumors, evolution and prognosis very variable.

The cytogenetic knowledge of DIA / DIG is very limited and is only available on small numbers of cases. Cytogenetic analyzes of several cases of DIG showed normal karyotypes. More recently, a CGH-Array study of 3 cases of DIA / DIG did not find any significant chromosomal gains or losses.

It has been shown, however, that a mutation involving BRAF (BRAF rearrangement or BRAF V600E mutations) was a recurrent element in low grade gliomas, particularly in pediatric patients.

It is also suggested that deregulation of BRAF activity in some DIA / DIG may indicate the importance of the MAPK (mitogen-activated protein kinase) pathway in signaling pathways for DIA / DIG development. However, data on the link between the BRAF gene and DIA / DIG remains very limited. Thus, further studies are needed to study the other members of the MAPK pathway in DIA / DIG (eg PI3K / AKT / mTOR). This could provide new therapeutic possibilities involving targeted therapies specific to the MAPK signaling pathway.

It appears that DIA / DIG does not all behave in a benign manner and some would undergo a malignant transformation that could be due to chromosomal alterations such as, for example, TP53, PI3K. In addition, because of the limited number of cases, it would be interesting to study the characteristics of patients with DIA / DIG in order to study their characteristics and whether there are clinical, pathological, cytogenetic and / Molecular forms between benign and malignant forms.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients,
* under the age of 18 at the time of diagnosis,
* carriers of a brain tumor diagnosed as a DIA or a DIG
* taken care of in a French referral center in pediatric oncology (centers of the French Society for Childhood Cancer, SFCE) between 01/01/1996 and 31/12/2015
* no reply to the newsletter

Exclusion Criteria:

* absence of pathologic confirmation of the diagnosis of DIA or DIG.
* absence of contact with one of the centers of the SFCE (a patient for whom an opinion on the conduct to be held before a DIA / DIG would have been requested from a reference service in pediatric oncology, may be included in the study. However, a record of this opinion must be present in the patient's medical record.)
* absence of fabric available

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with a brain tumor diagnosed as a DIA or DIG in a French referral center for pediatric oncology
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-08-18 (Actual); Primary Completion 2017-08-18 (Estimated); Study Completion 2017-08-18 (Estimated)

PRIMARY OUTCOMES:
Distribution of the characteristics of patients with DIA / DIG treated in the French SFCE pediatric oncology centers according to whether these tumors are benign or present a malignant transformation | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France